CLINICAL TRIAL: NCT03287063
Title: A Prospective Study Using Genomic, Histologic and Radiomic Analysis to Evaluate Regional Tumor Heterogeneity in Patients Undergoing Surgery for Newly Diagnosed Glioblastoma
Brief Title: Study Using Genomic, Histologic and Radiomic Analysis to Evaluate Regional Tumor Heterogeneity in Patients Undergoing Surgery for Newly Diagnosed Glioblastoma
Status: Terminated | Type: Observational
Why Stopped: Enrollment and/or interactions/interventions were halted prematurely due to loss of funding.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2017.094; HUM00134165 (Other: University of Michigan)
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be analyzed with next generation sequencing (NGS). The primary objective is to identify candidate genes with differential expression in therapy-resistant imaging subvolumes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tumor Biopsy — Stereotactic biopsies will be performed prior to resection.

SUMMARY:
Glioblastomas (GBM) demonstrate in vivo genetic and histologic heterogeneity that can be non-invasively identified using imaging phenotypes that identify regionally distinct areas of tumor with genetic alterations that drive tumor resistance pathways. The researchers propose a unique approach to assess initial GBM heterogeneity by performing histological and genomic analysis of biopsies targeted by advanced MRI before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Suspected newly diagnosed or recurrent supratentorial glioblastoma eligible for surgical biopsy and/or resection
* Patients must be 18 years of age or older
* Study-specific informed consent approved for this purpose by the IRB of the University of Michigan

Exclusion Criteria:

* Patients unable to undergo MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioblastoma eligible for surgical biopsy and/or resection
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Identify candidate genes with differential expression in therapy-resistant imaging subvolumes | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kim, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided